CLINICAL TRIAL: NCT02599701
Title: Acute Effects of Gabapentin on Polysomnography Parameters and on Hypothalamic-pituitary-adrenal, Hypothalamic-pituitary-gonadal and Somatotropic Axes During Sleep in Older Men: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Acute Effects of Gabapentin in Sleep Parameters and Hormonal Release During Sleep in Older Men
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Gabapentin increased hypopnea-apnea index in the first 8 recruited subjects.
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Dalva Poyares, Professor, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AFIP06/2015
Record Dates: First submitted 2015-07-21; First posted 2015-11-09 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Sleep
Keywords: Delta Sleep; Growth Hormone; IGF-1
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): A single dose of placebo with exactly the same characteristics of the active drug at bedtime.
  Interventions: Drug: Placebo
- Gabapentin (Experimental): A single dose of Gabapentin 300mg at bedtime.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — A single dose Gabapentin 300mg at bedtime.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo — A single placebo dose with the same physical characteristics of the active intervention.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effects of gabapentin in sleep polysomnography parameters and in nocturnal secretion of endogenous hypothalamic-pituitary-adrenal (HPA), hypothalamic-pituitary-gonadal (HPG) and somatotropic axes hormones and basal IGF-1 in older men.

DETAILED DESCRIPTION:
The influence of sleep variables on muscle protein anabolism is little studied, but data on the effects of slow-wave sleep and the syndrome of obstructive sleep apnea on the hypothalamic-pituitary axis indicate that interventions in the sleep structure and disorders impact on the age-related muscle loss. Thus, we propose to assess the acute effects of a drug potentially capable of increasing slow wave sleep, and consequently growth hormone release during sleep, on the physiological release of growth hormone, testosterone and IGF-1 during the night in older healthy men.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or more,
* healthy men

Exclusion Criteria:

* Basal Apnea-Hypopnea index (aHI)>=15
* Restless Legs Syndrome Symptons
* BMI less than 18.5 kg/m2 or greater than 30 kg/m2
* Less than 30 min. of regular physical activity (at least walking inside home, etc.)
* Plasma albumin below 3.5 mg/dL
* Psychoactive drugs use
* Drugs with muscle anabolic potential
* Current treatment for obesity or weight gain
* Enteral or parenteral feeding
* Inability to walk without assistance,
* Loss of independence in any activity of daily living
* Nocturia above 2 episodes
* Smoking more than 2 cigarettes per day
* Alcoholism (more than 2 doses a day)
* Prior epilepsy diagnosis
* Clinically evident atherosclerotic disease
* Dementia
* Depression
* Rheumatic diseases
* Cancer
* Diabetes (poorly controlled, HbA1C > 7,0, requirement of insulin)
* Thyroid dysfunction without treatment
* Advanced stages in COPD, HF, liver or renal failure

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Growth Hormone Secretion | During only one sleep night immediately after a single gabapentin or placebo dose at bedtime.
  Every 20 minutes after admission to the laboratory, blood samples (2.5 mL) for GH measurement will be collected (between 20:00 - or 2 hours before lights off - and 06:00).
IGF-1 | Immediately after the sleep night in that gabapentin or placebo dose were given at bedtime.
  It will be included in the analysis of the last sample collected for GH, testosterone and cortisol measurements at 06:00.

SECONDARY OUTCOMES:
Total testosterone | During only one sleep night immediately after a single gabapentin or placebo dose at bedtime.
  Every 20 minutes after admission to the laboratory, blood samples (2.5 mL) for free and total testosterone measurements will be collected (between 20:00 - or 2 hours before lights off - and 06:00).
Free testosterone | During only one sleep night immediately after a single gabapentin or placebo dose at bedtime.
  Every 20 minutes after admission to the laboratory, blood samples (2.5 mL) for free and total testosterone measurements will be collected (between 20:00 - or 2 hours before lights off - and 06:00).
Cortisol | During only one sleep night immediately after a single gabapentin or placebo dose at bedtime.
  Every 20 minutes after admission to the laboratory, blood samples (2.5 mL) for cortisol measurement will be collected (between 20:00 - or 2 hours before lights off - and 06:00).
Apnea-Hypopnea Index during sleep | During only one sleep night immediately after a single gabapentin or placebo dose at bedtime. a single gabapentin or placebo dose at bedtime.
  Sedative drugs may increase asymptomatic airway collapsability during sleep mainly in older individuals
Slow Wave Sleep - Stage N3 | During only one sleep night immediately after a single gabapentin or placebo dose at bedtime.
  Full sleep night polysomnographic recording.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Tufik, PhD, Study Chair — AFIP - Associação Fundo de Incentivo a Pesquisa
Locations (1):
- Instituto do Sono, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Giannoulis MG, Martin FC, Nair KS, Umpleby AM, Sonksen P. Hormone replacement therapy and physical function in healthy older men. Time to talk hormones? Endocr Rev. 2012 Jun;33(3):314-77. doi: 10.1210/er.2012-1002. Epub 2012 Mar 20. PMID 22433122
- [Background] Giustina A, Veldhuis JD. Pathophysiology of the neuroregulation of growth hormone secretion in experimental animals and the human. Endocr Rev. 1998 Dec;19(6):717-97. doi: 10.1210/edrv.19.6.0353. PMID 9861545
- [Background] Dattilo M, Antunes HK, Medeiros A, Monico Neto M, Souza HS, Tufik S, de Mello MT. Sleep and muscle recovery: endocrinological and molecular basis for a new and promising hypothesis. Med Hypotheses. 2011 Aug;77(2):220-2. doi: 10.1016/j.mehy.2011.04.017. Epub 2011 May 7. PMID 21550729
- [Background] Penev P, Spiegel K, L'Hermite-Baleriaux M, Schneider R, Van Cauter E. Relationship between REM sleep and testosterone secretion in older men. Ann Endocrinol (Paris). 2003 Apr;64(2):157. No abstract available. PMID 12773954
- [Background] Van Cauter E, Latta F, Nedeltcheva A, Spiegel K, Leproult R, Vandenbril C, Weiss R, Mockel J, Legros JJ, Copinschi G. Reciprocal interactions between the GH axis and sleep. Growth Horm IGF Res. 2004 Jun;14 Suppl A:S10-7. doi: 10.1016/j.ghir.2004.03.006. PMID 15135771
- [Background] Saletu M, Anderer P, Saletu-Zyhlarz GM, Parapatics S, Gruber G, Nia S, Saletu B. Comparative placebo-controlled polysomnographic and psychometric studies on the acute effects of gabapentin versus ropinirole in restless legs syndrome. J Neural Transm (Vienna). 2010 Apr;117(4):463-73. doi: 10.1007/s00702-009-0361-3. Epub 2010 Jan 5. PMID 20049491
- [Background] Foldvary-Schaefer N, De Leon Sanchez I, Karafa M, Mascha E, Dinner D, Morris HH. Gabapentin increases slow-wave sleep in normal adults. Epilepsia. 2002 Dec;43(12):1493-7. doi: 10.1046/j.1528-1157.2002.21002.x. PMID 12460250
- [Background] Rosenberg KP. Gabapentin for chronic insomnia. Am J Addict. 2003 May-Jun;12(3):273-4. No abstract available. PMID 12851024